CLINICAL TRIAL: NCT02791945
Title: N-acetylcysteine Treatment of Alcohol Use Disorder In Veterans With TBI
Acronym: NAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Northern California Institute of Research and Education (Other); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); Institute for Translational Neuroscience (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9236sc
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Traumatic Brain Injury (TBI); Hazardous and Harmful Alcohol Use
Keywords: TBI; hazardous and harmful alcohol use; Veterans; co-occurring disorders; pharmacotherapy
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetylcysteine (Experimental): N-acetylcysteine capsules daily - up to 3200 mg
  Interventions: Behavioral: Medical Management Counseling; Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Placebo capsules daily - up to 3200 mg
  Interventions: Behavioral: Medical Management Counseling; Drug: Placebo

INTERVENTIONS:
Behavioral: Medical Management Counseling — Brief alcohol counseling
Drug: N-acetylcysteine — Experimental supplement
  Other Names: NAC
  Arms: N-acetylcysteine
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
The goal of the project is to improve the care of Veterans with mild traumatic brain injury (mTBI) and unhealthy alcohol use.

DETAILED DESCRIPTION:
This is a pilot controlled clinical trial that aims to assess the efficacy of N-acetylcysteine (NAC) to reduce alcohol use and improve brain injury symptoms in Veterans with mTBI who consume alcohol at hazardous or harmful levels.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female veterans
2. Ages 18-65 (inclusive)
3. A history of mTBI as defined by American Congress of Rehabilitation Medicine (ACRM), in the chronic, stable phase of recovery (>6 months from injury).
4. Current (past month [30 days]) Hazardous or Harmful Alcohol Use: Hazardous use is drinking that meets NIAAA criteria: Current (past 30 day) weekly drinking, consisting of an average of 15 standard drinks/week for men or 8 standard drinks/week for women. Harmful use is drinking behavior that meets DSM-5 criteria mild AUD.
5. Participants must express a desire to reduce or stop alcohol use.
6. Female subjects that must have a negative urine pregnancy test and must be either postmenopausal one year or practicing an effective birth control method.

Exclusion Criteria:

1. Unstable psychotic or bipolar disorders, dementia, or other psychiatric disorders judged to be unstable in the clinical judgment of the PI or study physician.
2. Clinically significant unstable medical conditions, in the clinical judgment of the PI or study physician.
3. Female patients who are pregnant or nursing.
4. Concurrent participation in another alcohol treatment study, or in any research study involving medications.
5. Requiring acute medical detoxification from alcohol based on a score of 12 or more on the Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA-AD).
6. NAC use in the past week prior to study entry.
7. Use of AUD treatment medications (disulfiram, naltrexone, or acamprosate) within the past week.
8. Participants who are legally mandated to participate in an alcohol treatment program.
9. Participants who have had a suicide attempt in the past 3 months or suicidal ideation, with intent, in the 30 days prior to enrollment.
10. Participants who in the opinion of the investigator should not be enrolled in the study because of the precautions, warnings or contraindications outlined in the NAC package insert.
11. Participants with known hypersensitivity to acetylcysteine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Batki, MD, Principal Investigator — Unviersity of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-acetylcysteine | Placebo
Started | 14 | 16
Completed | 12 | 14
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine | Placebo | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49 (8) | 54 (10) | 52 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 12 | 16 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 6 | 8 | 14
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent of Heavy Drinking Days Per Week as Assessed by the Timeline Followback (TFLB)
Description: The TLFB interview, using a calendar, asks participants to report the prior week's frequency of alcohol use on each day of the week.
Time Frame: Baseline to Week 8
Measure: Mean (Standard Deviation); unit: change in percent heavy drinking days/wk
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 12 | 14
change in percent heavy drinking days/wk | 26.2 (0.31) | 26.5 (0.39)

2. Primary Outcome: Change in TBI Symptoms as Assessed by the Neurobehavioral Symptom Inventory (NSI)
Description: Participants indicate the extent to which each of the 22 symptoms has disturbed them in the previous 2 weeks on a 5-item scale (0-none to 4-severe). The NSI total score is the sum of severity ratings of the symptoms. The scores are summed to yield a total score ranging from 0 to 88, where the higher the point value, the greater (more severe) the symptoms
Time Frame: Baseline to Week 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 9 | 14
scores on a scale | 11.44 (10.09) | 10 (10.72)

3. Other Pre Specified Outcome: Change in Number of Standard Drinks Per Week as Assessed by the Timeline Followback (TLFB)
Description: as for outcome 1
Time Frame: Baseline to Week 8
Measure: Mean (Standard Deviation); unit: Standard drinks per week
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 12 | 14
Standard drinks per week | 24.75 (25.6) | 18.45 (30.1)

ADVERSE EVENTS:
Time Frame: Over 12 weeks.
Description: We used the Adverse Event Symptom Checklist at every study visit (Visits 0 - 8 and 12), which assessed the most reported adverse events listed in the FDA Prescribing Information.
Arm/Group | N-acetylcysteine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/16
Other Adverse Events (participants affected / at risk) | 14/14 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (N=14) | Placebo (N=16)
Inpatient hospitalization for self-reported "broken back in 3 places". (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Inpatient hospitalization/5150 (<72 hours) for suicidal threats while intoxicated (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (N=14) | Placebo (N=16)
Flushing (Skin and subcutaneous tissue disorders) | 1 | 4
Itching (Skin and subcutaneous tissue disorders) | 6 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 3
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 3
Nausea (Gastrointestinal disorders) | 0 (0) | 5
Vomiting (Gastrointestinal disorders) | 4 | 0
Upset stomach (Gastrointestinal disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT02791945/Prot_SAP_001.pdf
  • Informed Consent Form (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02791945/ICF_000.pdf